CLINICAL TRIAL: NCT04542070
Title: A Phase IIIb, Randomized, Multicenter, Active-controlled, Parallel-group, Non-inferiority, Open-label Study Evaluating the Efficacy, Safety, and Tolerability of Switching to Long-acting Cabotegravir Plus Long-acting Rilpivirine Administered Every Two Months From a Bictegravir/Emtricitabine/Tenofovir Alafenamide Single Tablet Regimen in HIV-1 Infected Adults Who Are Virologically Suppressed
Brief Title: A Study to Evaluate Efficacy and Safety of Cabotegravir (CAB) Long Acting (LA) Plus (+) Rilpivirine (RPV) LA Versus BIKTARVY® (BIK) in Participants With Human Immunodeficiency Virus (HIV)-1 Who Are Virologically Suppressed
Acronym: SOLAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 213500
Expanded Access: NCT03462810 (Available)
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: HIV Infections
Keywords: HIV; Cabotegravir; Rilpivirine; BIKTARVY; Antiretroviral therapy
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Rilpivirine; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Biktarvy (BIK) (Active Comparator): Participants with HIV-1 received BIK tablet orally until month 12. BIK was a fixed dose combination of 50 mg Bictegravir (BIC) + 200 mg Emtricitabine (FTC) + 25 mg Tenofovir alafenamide (TAF).
  Interventions: Drug: BIKTARVY Tablets (BIK)
- Oral lead-in phase (OLI) (Experimental): Participants with human immunodeficiency viruses (HIV)-1 who chose oral lead in (OLI) received oral 30 milligram (mg) Cabotegravir (CAB) tablet + 25 mg Rilpivirine (RPV) tablet once daily (QD) for one month. At the month 1 visit, the last dose of oral CAB + RPV was given, followed by the first 600 mg CAB long-acting (LA) + 900 mg RPV LA intramuscular injection (IM), and second injection of CAB LA 600 mg + RPV LA 900 mg at month 2, and then subsequent injections once every 2 months (Q2M) until Month 12 (Maintenance Phase). The participants had the option to continue the regimen in the Extension Phase
  Interventions: Drug: Cabotegravir Tablets; Drug: Rilpivirine Tablets
- Direct to injections (D2I) (Experimental): Participants with HIV-1 who chose direct to injections (D2I) received the first injections of 600 mg CAB LA + 900 mg RPV LA, IM as initial loading doses at Day 1 one month, followed by second and third subsequent injections (CAB LA 600 mg + RPV LA 900 mg) at month 1 and month 3 followed by Q2M until Month 11. The participants had the option to continue the regimen in the Extension Phase.
  Interventions: Drug: Cabotegravir Injectable Suspension (CAB LA); Drug: Rilpivirine Injectable Suspension (RPV LA)
- Switch Q2M Group (Active Comparator): Eligible participants with HIV-1 who received BIK tablet orally switched treatment after month 12 (Extension Phase) to CAB LA 600 mg + RPV LA 900 mg regimen, administered once every 2 months.
  Interventions: Drug: Cabotegravir Injectable Suspension (CAB LA); Drug: Rilpivirine Injectable Suspension (RPV LA)

INTERVENTIONS:
Drug: Cabotegravir Tablets — CAB tablets were available as film coated tablets for oral administration.
  Arms: Oral lead-in phase (OLI)
Drug: Cabotegravir Injectable Suspension (CAB LA) — CAB LA was available as sterile suspension for injection in GSK1265744 for administration as IM injection.
  Arms: Direct to injections (D2I); Switch Q2M Group
Drug: Rilpivirine Tablets — RPV was administered as tablets for oral administration.
  Arms: Oral lead-in phase (OLI)
Drug: Rilpivirine Injectable Suspension (RPV LA) — RPV LA was available as a sterile suspension of RPV to be administered as an IM injection.
  Arms: Direct to injections (D2I); Switch Q2M Group
Drug: BIKTARVY Tablets (BIK) — BIK was a three-drug fixed dose combination product BIC, FTC, and TAF for oral administration.
  Arms: Biktarvy (BIK)

SUMMARY:
This study is designed to assess the antiviral activity and safety of a two-drug regimen of CAB LA + RPV LA compared with maintenance of BIK. BIKTARVY is a registered trademark of Gilead Sciences.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older (or >=19 where required by local regulatory agencies), at the time of signing the informed consent.
* A female participant is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotropin (hCG) test at screen and a negative urine hCG test at Randomization), not lactating, and at least one of the following conditions applies.

  1. Non-reproductive potential defined as:

     * Pre-menopausal females with one of the following:

       1. Documented tubal ligation.
       2. Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion.
       3. Hysterectomy.
       4. Documented Bilateral Oophorectomy
     * Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.
  2. Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication, throughout the study, for at least 30 days after discontinuation of all oral study medications, and for at least 52 weeks after discontinuation of CAB LA and RPV LA.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in this protocol. Eligible participants or their legal guardians (and next of kin when locally required), must sign a written Informed Consent Form before any protocol-specified assessments are conducted. Enrollment of participants who are unable to provide direct informed consent is optional and will be based on local legal/regulatory requirements and site feasibility to conduct protocol procedures.
* Participants enrolled in France must be affiliated to, or a beneficiary of, a social security category.
* Must be on the uninterrupted current regimen of BIK for at least 6 months prior to Screening with an undetectable HIV-1 viral load for at least 6 months prior to Screening. BIK must be the participant's first or second regimen. If BIK is the second regimen, the first regimen must be an integrase inhibitor (INI) regimen. Only a single prior Integrase inhibitor (INI) regimen is allowed if BIK is a second line regimen >=6 months prior to screening. Any history of non-integrase strand transfer inhibitor regimens (that is. non-nucleoside reverse transcriptase inhibitor, protease inhibitor, C-C chemokine receptor 5 and other entry inhibitors) are not permitted. Any prior change in regimen, defined as a change of a single drug or multiple drugs simultaneously, must have occurred due to tolerability/safety, access to medications, or convenience/simplification, and must not have been done for treatment failure (HIV-1 RNA >=400 c/mL).

The following are limited exceptions:

* A change from Tenofovir disoproxil fumarate (TDF) to TAF will not be considered a regimen change.
* Historical perinatal use of Nucleoside reverse transcriptase inhibitor (NRTI) when given in addition to an ongoing Highly active antiretroviral therapy (HAART) will not be considered a change in ART therapy regimen.
* The past use of ARVs in the context of Post Exposure Prophylaxis (PEP) or Pre-Exposure Prophylaxis (PrEP) while the participant was HIV negative will be allowed. Such cases will be evaluated on a case by case basis with the Medical Monitor, and may require documentation of HIV negative serology during time of PEP or PrEP.
* A change in dosing scheme of the same drug from twice daily to once daily will not be considered a change in ART regimen if data support similar exposures and efficacy.
* A change in formulation from multiple class regimens to single treatment regimens (of the same medications) would not be considered a change in ART regimen.

  * Documented evidence of plasma HIV-1 RNA measurements <50 c/mL in the 6 months prior to Screening.
  * Plasma HIV-1 RNA <50 c/mL at Screening.

Exclusion Criteria:

* Within 6 months prior to Screening, any plasma HIV-1 RNA measurement >=50 c/mL.
* Within the 6 to 12-month window prior to Screening, documented evidence of any plasma HIV-1 RNA measurement greater than (>)200 c/mL, or 2 or more plasma HIV-1 RNA measurements >=50 c/mL.
* History of prior treatment failure to any Department of Health and Human Services (DHHS) recommended ART regimen.
* History of drug holiday >1 month for any reason prior to Screening visit, except where all ART was stopped due to tolerability and/or safety concerns.
* Any change to a second line regimen, defined as change of a single drug or multiple drugs simultaneously, due to virologic failure to therapy (defined as a confirmed plasma HIV 1 RNA measurement >=200 c/mL after initial suppression to <50 c/mL while on first line HIV therapy regimen).
* Participants who are currently participating in or anticipate being selected for any other interventional study.
* Women who are pregnant, breastfeeding or plan to become pregnant or breastfeed during the study.
* Any evidence of a current Center for Disease Control and Prevention (CDC) Stage 3 disease except cutaneous Kaposi's sarcoma not requiring systemic therapy, and CD4+ counts <200 cells/microliter are not exclusionary.
* Participants with moderate to severe hepatic impairment.
* Any pre-existing physical or mental condition (including substance use disorder) which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Participants determined by the Investigator to have a high risk of seizures, including participants with an unstable or poorly controlled seizure disorder. A participant with a prior history of seizure may be considered for enrollment if the Investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the Medical Monitor prior to enrollment.
* All participants will be screened for syphilis.

  * Participants with untreated secondary (late latent) or tertiary syphilis infection, defined as a positive rapid plasma reagin (RPR) and a positive treponemal test without clear documentation of treatment, are excluded.
  * Participants with a false positive RPR (with negative treponemal test) or serofast RPR result (persistence of a reactive nontreponemal syphilis test despite history of adequate therapy and no evidence of re-exposure) may enroll after consultation with the Medical Monitor.
  * Participants with primary syphilis or early latent secondary syphilis (acquired within the preceding year) who have a positive RPR test and have not been treated may be treated during the screening period and if completion of antibiotic treatment occurs during the screening period, may be allowed entry after consultation with the Medical Monitor. If antibiotic treatment cannot be completed before the screening window ends, participants may be rescreened once following completion of antibiotic therapy for primary or early latent secondary syphilis.
* Participants who, in the investigator's judgment, pose a significant suicide risk. Participant's recent history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.
* The participant has a tattoo, gluteal implant/enhancements or other dermatological condition overlying the gluteus region which may interfere with interpretation of injection site reactions.
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antibody (anti-HBs) and HBV deoxyribonucleic acid (DNA) as follows:

  1. Participants positive for HBsAg are excluded.
  2. Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status), whether negative or positive for HBV DNA, are excluded.
* Asymptomatic individuals with chronic hepatitis C virus (HCV) infection will not be excluded, however Investigators must carefully assess if therapy specific for HCV infection is required; participants who require or qualify for immediate HCV treatment are excluded for those co-infected participants who post entry into Switch Onto Long Acting Regimen (SOLAR) decide treatment for HCV infection is warranted or desired either by the participant or by the treating physician.

Participants with HCV co-infection will be allowed entry into this study if:

1. Liver enzymes meet entry criteria
2. HCV Disease has undergone appropriate work-up, and is not advanced, and will not require treatment prior to the Month 14 visit. Additional information (where available) on participants with HCV co-infection at screening should include results from any liver biopsy, Fibroscan, ultrasound, or other fibrosis evaluation, history of cirrhosis or other decompensated liver disease, prior treatment, and timing/plan for HCV treatment.
3. In the event that recent biopsy or imaging data is not available or inconclusive, the fibrosis (Fib)-4 score will be used to verify eligibility

i. Fib-4 score >3.25 is exclusionary ii. Fib-4 scores 1.45-3.25 requires Medical Monitor consultation Fibrosis 4 Score Formula: d. Age x aspartate aminotransferase (AST)/ Platelets x (square [Alanine aminotransferase {ALT}]).

* Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis, or decompensated cirrhosis [for example {e.g.} ascites, encephalopathy, or variceal bleeding]), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* History of liver cirrhosis with or without hepatitis viral co-infection.
* Ongoing or clinically relevant pancreatitis
* Clinically significant cardiovascular disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the participant prior to randomization.
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive study medication.
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class. In addition, if heparin is used during pharmacokinetic (PK) sampling, participants with a history of sensitivity to heparin or heparin-induced thrombocytopenia must not be enrolled.
* Current or anticipated need for chronic anti-coagulation with the exception of the use of low dose acetylsalicylic acid (less than or equal to [<=]325 milligram) or hereditary coagulation and platelet disorders such as hemophilia or Von Willebrand Disease.
* Corrected QT interval (QTc [Bazett]) >450 milliseconds (msec) or QTc (Bazett) >480 msec for participants with bundle branch block.
* Known or suspected active Coronavirus Disease-2019 (COVID-19) infection or has had contact with an individual with known COVID-19, within 14 days of study enrollment.
* Known or suspected presence of resistance mutations as defined by the International Antiviral Society-United States of America (IAS-USA) resistance guidelines to the individual components of BIK (BIC, FTC, TAF), RPV, and CAB by any historical resistance test result.
* Any verified Grade 4 laboratory abnormality. A single repeat test is allowed during the Screening phase to verify a result.
* Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the participant's participation in the study of an investigational compound.
* Participant has estimated creatine clearance <30mL/minute per 1.73 meter square (m^2) via Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) Method.
* ALT >=3 times upper limit of normal (ULN).
* Exposure to an experimental drug or experimental vaccine within either 30 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to Day 1 of this study.
* Treatment with any of the following agents within 28 days of Screening:

  * radiation therapy;
  * cytotoxic chemotherapeutic agents;
  * tuberculosis therapy with the exception of isoniazid (isonicotinylhydrazid/INH);
  * anti-coagulation agents;
  * Immunomodulators that alter immune responses such as chronic systemic corticosteroids, interleukins, or interferons.
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
* Treatment with any agent, except recognized ART as allowed above, with documented activity against HIV-1 within 28 days of study Day 1. Treatment with acyclovir/valacyclovir is permitted.
* Use of medications which are associated with Torsade de Pointes.
* Participants receiving any prohibited medication and who are unwilling or unable to switch to an alternate medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 687 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (95):
- United States (35):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Huntersville, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- Australia (4):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Darlinghurst, Sydney, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Prahran, Victoria
- Austria (3):
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Vienna
- Belgium (4):
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Lodelinsart
- Canada (5):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
- France (8):
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Tourcoing
- Germany (7):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Dublin, Ireland
- Italy (8):
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Busto Arsizio (VA), Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Turin, Piedmont
- Japan (3):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Amsterdam, Netherlands
- Spain (8):
  - GSK Investigational Site, Alcalá de Henares
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Huelva
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda( Madrid
  - GSK Investigational Site, Sant Boi de Llobregat
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Switzerland (4):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Geneva
  - GSK Investigational Site, Lausanne
  - GSK Investigational Site, Zurich
- United Kingdom (4):
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on ViiV's data sharing criteria can be found at: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/

REFERENCES:
- [Background] Karver TS, Pascual-Bernaldez M, Berni A, Hnoosh A, Castagna A, Messiaen P, Puerto MJG, Bloch M, Adachi E, Sinclair G, Felizarta F, Angel JB, Sutton K, Sutherland-Phillips D, D'Amico R, Kerrigan D. Factors Associated with Health Care Providers' Preference for Forgoing an Oral Lead-In Phase When Initiating Long-Acting Injectable Cabotegravir and Rilpivirine in the SOLAR Clinical Trial. AIDS Patient Care STDS. 2023 Jan;37(1):53-59. doi: 10.1089/apc.2022.0168. PMID 36626155
- [Background] Ramgopal MN, Castagna A, Cazanave C, Diaz-Brito V, Dretler R, Oka S, Osiyemi O, Walmsley S, Sims J, Di Perri G, Sutton K, Sutherland-Phillips D, Berni A, Latham CL, Zhang F, D'Amico R, Pascual Bernaldez M, Van Solingen-Ristea R, Van Eygen V, Patel P, Chounta V, Spreen WR, Garges HP, Smith K, van Wyk J. Efficacy, safety, and tolerability of switching to long-acting cabotegravir plus rilpivirine versus continuing fixed-dose bictegravir, emtricitabine, and tenofovir alafenamide in virologically suppressed adults with HIV, 12-month results (SOLAR): a randomised, open-label, phase 3b, non-inferiority trial. Lancet HIV. 2023 Sep;10(9):e566-e577. doi: 10.1016/S2352-3018(23)00136-4. Epub 2023 Aug 8. PMID 37567205
- [Derived] Adachi E, Yokomaku Y, Watanabe D, Gatanaga H, Oka S, Shirasaka T, D'Amico R, Sutton K, Sutherland-Phillips D, Roberts J, Thornhill J, Murungi A, Brown K. Month 12 outcomes of switching to long-acting cabotegravir + rilpivirine with an oral lead-in versus continuing bictegravir/emtricitabine/tenofovir alafenamide in the Phase 3b randomized SOLAR study. J Infect Chemother. 2025 Dec;31(12):102834. doi: 10.1016/j.jiac.2025.102834. Epub 2025 Oct 17. PMID 41110828
- [Derived] Adachi E, Yokomaku Y, Watanabe D, Gatanaga H, Oka S, Shirasaka T, Wakatabe R, Chamay N, Sutton K, Sutherland-Phillips D, Urbaityte R, D'Amico R, van Wyk J. Efficacy and safety of switching to long-acting cabotegravir + rilpivirine versus continuing bictegravir/emtricitabine/tenofovir alafenamide in Japanese participants: 12-month results from the phase 3b randomized SOLAR trial. J Infect Chemother. 2025 Jul;31(7):102734. doi: 10.1016/j.jiac.2025.102734. Epub 2025 May 16. PMID 40383512
- [Derived] Tan DHS, Antinori A, Eu B, Galindo Puerto MJ, Kinder C, Sweet D, Van Dam CN, Sutton K, Sutherland-Phillips D, Berni A, Zhang F, Urbaityte R, Baugh B, Spreen W, van Wyk J, Garges HP, Patel P, Batterham R, D'Amico R. Weight and Metabolic Changes With Long-Acting Cabotegravir and Rilpivirine or Bictegravir/Emtricitabine/Tenofovir Alafenamide. J Acquir Immune Defic Syndr. 2025 Apr 1;98(4):401-409. doi: 10.1097/QAI.0000000000003584. Epub 2025 Feb 19. PMID 39676239

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consists in 2 periods: Maintenance Period and Extension Period. Any participants who successfully completed 12 months of CAB+RPV treatment in the Maintenance Phase had the option to enter the Extension Phase and continued to have access to CAB + RPV.
Pre-assignment Details: 687 participants were enrolled in this study, out of which 681 were included in intent-to-treat exposed population (ITT-E).The Modified ITT-E (excluded participants due to eligibility criteria violations and GCP non-compliance) was used to primarily present the participant flow, baseline characteristics and efficacy analysis. Safety analyses were primarily presented based on Safety set, which included all participants including the ones with eligibility criteria violations and GCP non-compliance
Period: Maintenance Period (Day 1 - Month 12)
Arm/Group | Oral lead-in Phase (OLI) | Direct to Injections (D2I) | Biktarvy (BIK) | Switch Q2M Group
Started (Intent-to-Treat-Exposed (ITT-E)) | 175 | 279 | 227 | 0 (Participants were transitioned to the Switch Q2M Group (from BIK regiment to CAB LA 600 mg + RPV LA 900 mg regimen) at the beginning of Extension Phase (Month 13).)
Completed | 152 | 255 | 213 | 0 (Participants were transitioned to the Switch Q2M Group (from BIK regiment to CAB LA 600 mg + RPV LA 900 mg regimen) at the beginning of Extension Phase (Month 13).)
Not Completed | 23 | 24 | 14 | 0
Not completed — Adverse Event | 10 | 3 | 1 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0 | 0
Not completed — Lost to Follow-up | 3 | 4 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 8 | 9 | 0
Not completed — Protocol Deviation | 2 | 6 | 1 | 0
Not completed — Protocol-Specified Withdrawal Criterion Met | 1 | 1 | 0 | 0
Period: Maintenance + Extension Period
Arm/Group | Oral lead-in Phase (OLI) | Direct to Injections (D2I) | Biktarvy (BIK) | Switch Q2M Group
Started | 173 (The participants in Oral lead-in phase (OLI) group received same treatment regimen in both Maintenance and Extension Phases, hence data was summarized by Maintenance Phase and by Maintenance+Extension Phase.) | 274 (The participants in Direct to injections (D2I) group received same treatment regimen in both Maintenance and Extension Phases, hence data was summarized by Maintenance Phase and by Maintenance+Extension Phase.) | 0 (Participants were transitioned to the Switch Q2M Group (from BIK regiment to CAB LA 600 mg + RPV LA 900 mg regimen) at the beginning of Extension Phase (Month 13), hence data was summarized by Maintenance Phase and by Extension Phase.) | 0 (Participants were transitioned to the Switch Q2M Group (from BIK regiment to CAB LA 600 mg + RPV LA 900 mg regimen) at the beginning of Extension Phase (Month 13).)
Completed | 150 | 247 | 0 (Participants were transitioned to the Switch Q2M Group (from BIK regiment to CAB LA 600 mg + RPV LA 900 mg regimen) at the beginning of Extension Phase (Month 13), hence data was summarized by Maintenance Phase and by Extension Phase.) | 0 (Participants were transitioned to the Switch Q2M Group (from BIK regiment to CAB LA 600 mg + RPV LA 900 mg regimen) at the beginning of Extension Phase (Month 13).)
Not Completed | 23 | 27 | 0 | 0
Not completed — Adverse Event | 10 | 2 | 0 | 0
Not completed — Lack of Efficacy | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 3 | 4 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 5 | 0 | 0
Not completed — Protocol-specified withdrawal criterion met | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 12 | 0 | 0
Period: Extension Period (Month 13 - Month 27)
Arm/Group | Oral lead-in Phase (OLI) | Direct to Injections (D2I) | Biktarvy (BIK) | Switch Q2M Group
Started | 0 (The participants in Oral lead-in phase (OLI) group received same treatment regimen in both Maintenance and Extension Phases, hence data was summarized by Maintenance Phase and by Maintenance+Extension Phase.) | 0 (The participants in Direct to injections (D2I) group received same treatment regimen in both Maintenance and Extension Phases, hence data was summarized by Maintenance Phase and by Maintenance+Extension Phase.) | 0 (Biktarvy (BIK) group was dissolved at the start of Extension Phase, when participants transitioned to Switch Q2M Group or commercial available treatments, based on protocol criteria.) | 143 (143 participants from the Biktarvy (BIK) group were eligible to transition to Switch Q2M Group at the start of Extension Phase.)
Completed | 0 | 0 | 0 | 130
Not Completed | 0 | 0 | 0 | 13
Not completed — Adverse Event | 0 | 0 | 0 | 4
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral lead-in Phase (OLI) | Direct to Injections (D2I) | Biktarvy (BIK) | Total
Number analyzed (Participants) | 175 | 279 | 227 | 681
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 38.5 (11.38) | 39.0 (11.09) | 38.6 (11.41) | 38.7 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 52 | 41 | 120
  Male | 148 | 227 | 186 | 561
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 4 | 2 | 16
  Asian - Central/South Asian Heritage | 0 | 3 | 0 | 3
  Asian - East Asian Heritage | 1 | 0 | 2 | 3
  Asian - Japanese Heritage | 4 | 10 | 6 | 20
  Asian - South East Asian Heritage | 2 | 3 | 3 | 8
  Black or African American | 40 | 56 | 49 | 145
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  White - Arabic/North African Heritage | 10 | 5 | 10 | 25
  White - White/Caucasian/European Heritage | 104 | 194 | 149 | 447
  Mixed White Race | 0 | 0 | 1 | 1
  Multiple | 4 | 4 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Viruses (HIV)-1 Ribonucleic Acid (RNA) Greater Than or Equal to (>=) 50 Copies Per Milliliter (c/mL) at Month 12/11 - ITT-E Population
Description: Percentage of participants with plasma HIV 1 RNA >= 50 c/mL at month 12 was assessed using the food and drug administration (FDA) snapshot algorithm. For the Q2M arm, data from the Q2M OLI participants at Month 12 visit and Q2M D2I participants at Month 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 12 visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit. The FDA snapshot algorithm defines a participant's virologic response status using only the viral load at the predefined time point within a window of time (HIV-RNA equal to or above 50 copies/mL and HIV-RNA below 50 copies/mL), along with study drug discontinuation status. The third category of the FDA snapshot ("No virologic data") is not pre-defined as an endpoint and therefore not reported separately.
Time Frame: At month 12/11
Population: Intent-to-treat exposed (ITT-E) population included all randomized participants who receive at least one dose of IP during the Maintenance Phase of the study (on or after Day 1).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Q2M (OLI + D2I): Participants with HIV-1 who started OLI were administered with Cabotegravir and Rilpivirine (CAB + RPV) tablets orally for one month. At the month 1 visit, the last dose of oral 30 mg CAB + 25 mg RPV tablets were given, followed by the first 600 mg CAB LA + 900 mg RPV LA intramuscular injection, and second injection of CAB LA 600 mg + RPV LA 900 mg at month 2, and then subsequent injections every 2 months (Q2M) until Month 12. Participants with HIV-1 who started with D2I, received the first injection of 600 mg CAB LA + 900 mg RPV LA, IM as initial loading dose at Day 1 followed by second and third subsequent injections (CAB LA 600 mg + RPV LA 900 mg) at month 1 and 3 followed by Q2M until Month 11.
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 454 | 227
Percentage of participants | 1.3 [0.5 to 2.9] | 0.4 [0.0 to 2.4]
Statistical Analysis 1: Comparison: Q2M (OLI + D2I) vs Biktarvy (BIK); Test type: Non-Inferiority — Non-inferiority concluded if the upper limit of a two-sided 95% confidence interval for the difference in percentage of participants with HIV-1 RNA ≥ 50 c/mL at Month 12 (OLI and BIK)/Month 11 (D2I) between the two treatment arms (Q2M - BIK) is less than 4%; Difference in percentage = 0.9, 95% CI 2-sided [-0.5 to 2.2] — Difference in percentage = percentage of Q2M - percentage of BIK
Statistical Analysis 2: Comparison: Q2M (OLI + D2I) vs Biktarvy (BIK); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Adjusted difference in percentage = 0.9, 95% CI 2-sided [-0.5 to 2.2] — Adjusted difference in percentage = percentage of Q2M - percentage of BIK. Based on cochran-mantel haenszel stratified analysis was adjusted for the baseline stratification factors gender at birth and baseline BMI

2. Primary Outcome: Percentage of Participants With Plasma HIV-1 RNA Greater >=50 Copies Per Milliliter (c/mL) at Month 12/11 - mITT-E Population
Description: as for outcome 1
Time Frame: At month 12/11
Population: Modified intent-to-treat exposed (mITT-E) population included all ITT-E participants (that is all randomized participants who received at least one dose of IP during the Maintenance Phase of the study [(on or after Day 1])) excluding those from a GSK Investigational site where Good Clinical Practice noncompliance was observed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 447 | 223
Percentage of participants | 1.1 [0.4 to 2.6] | 0.4 [0.0 to 2.5]
Statistical Analysis 1: Comparison: Q2M (OLI + D2I) vs Biktarvy (BIK); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in percentage = 0.7, 95% CI 2-sided [-0.6 to 2.0] — Difference in percentage = percentage of Q2M - percentage of BIK
Statistical Analysis 2: Comparison: Q2M (OLI + D2I) vs Biktarvy (BIK); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Adjusted difference in percentage = 0.7, 95% CI 2-sided [-0.7 to 2.0] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Less Than (<)50 c/mL at Month 12/11 - ITT-E Population
Description: Percentage of participants with plasma HIV 1 RNA < 50 c/mL was assessed using the FDA snapshot algorithm. For the Q2M arm, data from the Q2M OLI participants at Month 12 visit and Q2M D2I participants at Month 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 12 visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit. The FDA snapshot algorithm defines a participant's virologic response status using only the viral load at the predefined time point within a window of time (HIV-RNA equal to or above 50 copies/mL and HIV-RNA below 50 copies/mL), along with study drug discontinuation status. The third category of the FDA snapshot ("No virologic data") is not pre-defined as an endpoint and therefore not reported separately.
Time Frame: At month 12/11
Population: Intent-to-treat exposed (ITT-E) population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 454 | 227
Percentage of participants | 89.4 [86.6 to 92.3] | 93.0 [89.6 to 96.3]

4. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Month 12/11 -mITT-E Population
Description: as for outcome 3
Time Frame: At month 12/11
Population: Modified intent-to-treat exposed (mITT-E) population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 447 | 223
Percentage of participants | 90.2 [87.4 to 92.9] | 92.8 [89.4 to 96.2]

5. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Month 6/5 - ITT-E Population
Description: Percentage of participants with plasma HIV 1 RNA < 50 c/mL was assessed using the FDA snapshot algorithm. For the Q2M arm, data from the Q2M OLI participants at Month 6 visit and Q2M D2I participants at Month 5 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. The FDA snapshot algorithm defines a participant's virologic response status using only the viral load at the predefined time point within a window of time (HIV-RNA equal to or above 50 copies/mL and HIV-RNA below 50 copies/mL), along with study drug discontinuation status. The third category of the FDA snapshot ("No virologic data") is not pre-defined as an endpoint and therefore not reported separately.
Time Frame: At month 6/5
Population: Intent-to-treat exposed (ITT-E) population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 454 | 227
Percentage of participants | 92.7 [90.3 to 95.1] | 97.8 [95.9 to 99.7]

6. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Month 6/5 - mITT-E Population
Description: as for outcome 5
Time Frame: At month 6/5
Population: Modified intent-to-treat exposed (mITT-E) population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 447 | 223
Percentage of participants | 93.5 [91.2 to 95.8] | 97.8 [95.8 to 99.7]

7. Secondary Outcome: Number of Participants With Protocol-defined Confirmed Virologic Failure (CVF) Through Month 6/5 and 12/11
Description: Protocol-defined confirmed virologic failure was defined as rebound as indicated by two consecutive plasma HIV-1 RNA levels >= 200 c/mL (Day 1 values are not applicable) after prior suppression to <200 c/mL. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at Month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit. Cumulative number of participants with protocol defined CVF through Month 6/5 and 12/11 has been presented.
Time Frame: Up to month 12
Population: Modified intent-to-treat exposed (mITT-E) population
Measure: Count of Participants; unit: Participants
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 447 | 223
Participants
  Month 6/5 | 1 | 0
  Month 12/11 | 2 | 0

8. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA Greater Than or Equal to (>=) 50 c/mL at Month 6/5
Description: Percentage of participants with plasma HIV 1 RNA >= 50 c/mL at month 6 was assessed using the food and drug administration (FDA) snapshot algorithm. For the Q2M arm, data from the Q2M OLI participants at Month 6 visit and Q2M D2I participants at Month 5 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. The FDA snapshot algorithm defines a participant's virologic response status using only the viral load at the predefined time point within a window of time (HIV-RNA equal to or above 50 copies/mL and HIV-RNA below 50 copies/mL), along with study drug discontinuation status. The third category of the FDA snapshot ("No virologic data") is not pre-defined as an endpoint and therefore not reported separately.
Time Frame: At month 6/5
Population: Modified intent-to-treat exposed (mITT-E) population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 447 | 223
Percentage of participants | 0.4 [0.1 to 1.6] | 0 [0.0 to 1.6]

9. Secondary Outcome: Absolute Values of HIV Viral Load
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Logarithm to base 10 (log10) values for plasma HIV-1 RNA has been presented. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: Modified intent-to-treat exposed (mITT-E) population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: log10 copies per milliliter(c/mL)
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 447 | 223
log10 copies per milliliter(c/mL)
  Baseline (Day 1) | 1.5993 (0.10559) | 1.5947 (0.06640)
  Month 6/5: number analyzed (Participants) | 420 | 218
  Month 6/5 | 1.6002 (0.09268) | 1.5910 (0.01182)
  Month 12/11: number analyzed (Participants) | 406 | 201
  Month 12/11 | 1.6019 (0.13064) | 1.5911 (0.01552)

10. Secondary Outcome: Change From Baseline in HIV Viral Load
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is defined as post-dose visit value minus Baseline value. Logarithm to base 10 values for plasma HIV-1 RNA has been presented. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: log10 c/mL
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 447 | 223
log10 c/mL
  Baseline (Day 1) | 1.5993 (0.10559) | 1.5947 (0.06640)
  Month 6/5: number analyzed (Participants) | 420 | 218
  Month 6/5 | 0.0015 (0.13997) | -0.0039 (0.06826)
  Month 12/11: number analyzed (Participants) | 406 | 201
  Month 12/11 | 0.0029 (0.17038) | -0.0041 (0.07172)

11. Secondary Outcome: Absolute Values of Cluster of Differentiation 4 Plus (CD4+) Cell Count
Description: Blood samples were collected and CD4+ cell count was assessed using flow cytometry. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter(cells/mm^3)
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 447 | 222
cells per cubic millimeter(cells/mm^3)
  Baseline (Day 1) | 670.9 (282.11) | 679.4 (306.89)
  Month 6/5: number analyzed (Participants) | 412 | 212
  Month 6/5 | 689.1 (284.89) | 673.7 (290.46)
  Month 12/11: number analyzed (Participants) | 395 | 192
  Month 12/11 | 711.9 (297.13) | 717.3 (317.82)

12. Secondary Outcome: Change From Baseline in CD4+ Cell Count
Description: Blood samples were collected and CD4+ cell count was assessed using flow cytometry. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 447 | 223
cells/mm^3
  Baseline (Day 1) | 670.9 (282.11) | 679.4 (306.89)
  Month 6/5: number analyzed (Participants) | 412 | 211
  Month 6/5 | 20.4 (202.38) | -3.1 (197.62)
  Month 12/11: number analyzed (Participants) | 395 | 191
  Month 12/11 | 35.2 (219.79) | 32.2 (208.29)

13. Secondary Outcome: Number of Participants With Treatment-emergent Phenotypic Resistance Through Month 12/11
Description: Blood samples were collected to evaluate the phenotypic resistance to CAB, RPV, BIC, FTC, and TAF. For each participant, prevalence of phenotype, fold changes to CAB, RPV, and BIC, replication capacity of Integrase, protease, and reverse transcriptase enzymes at the time of CVF was assessed. For the Q2M arm, data from the Q2M OLI participants at Month 12 visit and Q2M D2I participants at Month 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 12 visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit. No participants in the BIK arm met CVF.
Time Frame: Up to Month 12/11
Population: Confirmed Virologic Failure (CVF) population included all participants in the ITT-E population who met Confirmed Virologic Failure (CVF).
Measure: Count of Participants; unit: Participants
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 2 | 0
Participants
  NNRTI | 2 | 0
  IN | 2 | 0

14. Secondary Outcome: Number of Participants With Treatment-emergent Phenotypic Resistance Through Month 6/5
Description: Blood samples were collected to evaluate the phenotypic resistance to CAB, RPV, BIC, FTC, and TAF. For each participant, prevalence of phenotype, fold changes to CAB, RPV, and BIC, replication capacity of Integrase, protease, and reverse transcriptase enzymes at the time of CVF was assessed. For the Q2M arm, data from the Q2M OLI participants at Month 6 visit and Q2M D2I participants at Month 5 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. No participants in the BIK arm met CVF.
Time Frame: Up to Month 6/5
Population: Confirmed Virologic Failure (CVF) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 1 | 0
Participants
  NNRTI | 1 | 0
  IN | 1 | 0

15. Secondary Outcome: Number of Participants With Treatment-emergent Genotypic Resistance Through Month 12/11
Description: Blood samples were collected to evaluate the genotypic resistance to CAB, RPV, BIC, FTC, and TAF. For each participant, prevalence of resistance mutations and genotypic susceptibility at the time of CVF was assessed. For the Q2M arm, data from the Q2M OLI participants at Month 12 visit and Q2M D2I participants at Month 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 12 visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit. No participants in the BIK arm met CVF.
Time Frame: Up to Month 12/11
Population: Confirmed Virologic Failure (CVF) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 2 | 0
Participants
  M230L | 1 | 0
  Q148R | 1 | 0
  K101E | 1 | 0
  G118R | 1 | 0

16. Secondary Outcome: Number of Participants With Treatment-emergent Genotypic Resistance Through Month 6/5
Description: Blood samples were collected to evaluate the genotypic resistance to CAB, RPV, BIC, FTC, and TAF. For each participant, prevalence of resistance mutations and genotypic susceptibility at the time of CVF was assessed. For the Q2M arm, data from the Q2M OLI participants at Month 6 visit and Q2M D2I participants at Month 5 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. No participants in the BIK arm met CVF.
Time Frame: Up to Month 6/5
Population: Confirmed Virologic Failure (CVF) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 1 | 0
Participants
  M230L | 1 | 0
  Q148R | 1 | 0

17. Secondary Outcome: Change From Baseline in Bone Biomarkers: Specific Alkaline Phosphatase, Procollagen Type 1 N-Terminal Propeptide, Type 1 Collagen Cross-linked C-telopeptide, Osteocalcin (Micrograms Per Liter (ug/L))
Description: Serum samples were collected to evaluate bone specific biomarkers: specific alkaline phosphatase, procollagen type 1 N-propeptide, type 1 collagen cross-linked C-telopeptide, osteocalcin. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: Safety Population included all randomly assigned participants who received at least one dose of study drug. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: micrograms per liter (ug/L)
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 449 | 227
micrograms per liter (ug/L)
  Serum Bone Specific Alkaline Phosphatase, Baseline (Day 1): number analyzed (Participants) | 448 | 227
  Serum Bone Specific Alkaline Phosphatase, Baseline (Day 1) | 12.7 (4.27) | 12.9 (4.60)
  Serum Bone Specific Alkaline Phosphatase, Month 6/5: number analyzed (Participants) | 418 | 221
  Serum Bone Specific Alkaline Phosphatase, Month 6/5 | 0.3 (9.89) | 0.2 (2.60)
  Serum Bone Specific Alkaline Phosphatase, Month 12/11: number analyzed (Participants) | 403 | 208
  Serum Bone Specific Alkaline Phosphatase, Month 12/11 | 0.1 (5.03) | 0.5 (3.55)
  Serum Osteocalcin, Baseline (Day 1): number analyzed (Participants) | 447 | 227
  Serum Osteocalcin, Baseline (Day 1) | 21.0 (7.35) | 20.4 (7.48)
  Serum Osteocalcin, Month 6/5: number analyzed (Participants) | 418 | 219
  Serum Osteocalcin, Month 6/5 | 0.4 (5.53) | -0.4 (5.11)
  Serum Osteocalcin, Month 12/11: number analyzed (Participants) | 395 | 209
  Serum Osteocalcin, Month 12/11 | 0.9 (6.11) | -0.6 (5.51)
  Serum Procollagen 1 N-Terminal Propeptide, Baseline (Day 1): number analyzed (Participants) | 448 | 226
  Serum Procollagen 1 N-Terminal Propeptide, Baseline (Day 1) | 59.1 (23.06) | 59.2 (23.88)
  Serum Procollagen 1 N-Terminal Propeptide, Month 6/5: number analyzed (Participants) | 420 | 219
  Serum Procollagen 1 N-Terminal Propeptide, Month 6/5 | -1.5 (15.70) | 0.1 (18.53)
  Serum Procollagen 1 N-Terminal Propeptide, Month 12/11: number analyzed (Participants) | 402 | 209
  Serum Procollagen 1 N-Terminal Propeptide, Month 12/11 | -0.7 (19.73) | 0.6 (19.63)
  Serum Type I Collagen C-Telopeptides, Baseline (Day 1): number analyzed (Participants) | 449 | 226
  Serum Type I Collagen C-Telopeptides, Baseline (Day 1) | 0.4 (0.25) | 0.5 (0.25)
  Serum Type I Collagen C-Telopeptides, Month 6/5: number analyzed (Participants) | 421 | 222
  Serum Type I Collagen C-Telopeptides, Month 6/5 | -0.1 (0.23) | -0.1 (0.21)
  Serum Type I Collagen C-Telopeptides, Month 12/11: number analyzed (Participants) | 405 | 209
  Serum Type I Collagen C-Telopeptides, Month 12/11 | 0.0 (0.25) | 0.0 (0.22)

18. Secondary Outcome: Change From Baseline in Bone Biomarkers: Serum 25-hydroxyvitamin D (Nanomoles Per Liter (Nmol/L))
Description: Serum samples were collected to evaluate bone specific biomarkers: serum 25-hydroxyvitamin D. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 440 | 219
nanomoles per liter (nmol/L)
  Baseline (Day 1) | 61.0 (34.69) | 59.9 (33.30)
  Month 6/5: number analyzed (Participants) | 403 | 214
  Month 6/5 | 2.8 (29.24) | 6.0 (34.16)
  Month 12/11: number analyzed (Participants) | 393 | 199
  Month 12/11 | -2.3 (29.00) | -3.1 (26.38)

19. Secondary Outcome: Change From Baseline in Renal Biomarkers: Specific Serum Beta-2 Microglobulin, Cystatin c, Retinol Binding Protein, Urine Beta-2 Microglobulin (Milligrams Per Liter [mg/L])
Description: Serum samples were collected to evaluate renal specific biomarkers: specific serum beta-2 microglobulin, cystatin c, retinol binding protein, urine beta-2 microglobulin. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 448 | 227
milligrams per liter (mg/L)
  Serum beta-2 microglobulin, Baseline (Day 1): number analyzed (Participants) | 447 | 227
  Serum beta-2 microglobulin, Baseline (Day 1) | 1.8 (0.40) | 1.8 (0.38)
  Serum beta-2 microglobulin, Month 6/5: number analyzed (Participants) | 413 | 223
  Serum beta-2 microglobulin, Month 6/5 | 0.0 (0.28) | 0.0 (0.28)
  Serum beta-2 microglobulin, Month 12/11: number analyzed (Participants) | 402 | 208
  Serum beta-2 microglobulin, Month 12/11 | 0.0 (0.33) | 0.0 (0.32)
  Serum cystatin C, Baseline (Day 1) | 0.9 (0.13) | 0.9 (0.14)
  Serum cystatin C, Month 6/5: number analyzed (Participants) | 416 | 223
  Serum cystatin C, Month 6/5 | 0.0 (0.08) | 0.0 (0.08)
  Serum cystatin C, Month 12/11: number analyzed (Participants) | 404 | 209
  Serum cystatin C, Month 12/11 | 0.0 (0.08) | 0.0 (0.08)
  Serum retinol binding protein, Baseline (Day 1): number analyzed (Participants) | 446 | 227
  Serum retinol binding protein, Baseline (Day 1) | 51.3 (13.01) | 52.2 (12.61)
  Serum retinol binding protein, Month 6/5: number analyzed (Participants) | 417 | 220
  Serum retinol binding protein, Month 6/5 | -1.0 (9.00) | -0.3 (8.75)
  Serum retinol binding protein, Month 12/11: number analyzed (Participants) | 397 | 208
  Serum retinol binding protein, Month 12/11 | -1.2 (9.24) | 0.2 (9.06)
  Urine beta-2 microglobulin, Baseline (Day 1): number analyzed (Participants) | 257 | 128
  Urine beta-2 microglobulin, Baseline (Day 1) | 0.2 (0.34) | 0.2 (0.40)
  Urine beta-2 microglobulin, Month 6/5: number analyzed (Participants) | 175 | 84
  Urine beta-2 microglobulin, Month 6/5 | 0.0 (0.40) | 0.1 (0.65)
  Urine beta-2 microglobulin, Month 12/11: number analyzed (Participants) | 148 | 86
  Urine beta-2 microglobulin, Month 12/11 | 0.0 (0.24) | 0.1 (0.52)

20. Secondary Outcome: Change From Baseline in Renal Biomarkers: Urine Phosphate (Millimoles Per Liter (mmol/L))
Description: Serum samples were collected to evaluate renal specific biomarkers: urine phosphate. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 449 | 223
millimoles per liter (mmol/L)
  Baseline (Day 1) | 20.0 (14.03) | 18.4 (13.10)
  Month 6/5: number analyzed (Participants) | 414 | 218
  Month 6/5 | -1.0 (16.29) | 0.4 (15.60)
  Month 12/11: number analyzed (Participants) | 399 | 205
  Month 12/11 | 0.1 (16.17) | -0.6 (15.16)

21. Secondary Outcome: Change From Baseline in Renal Biomarker: Urine Retinol Binding Protein 4 (Microgram Per Liter (ug/L))
Description: Serum samples were collected to evaluate renal specific biomarkers: urine retinol binding protein 4. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: microgram per liter (ug/L)
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 447 | 222
microgram per liter (ug/L)
  Baseline (Day 1) | 114.2 (111.45) | 100.0 (82.00)
  Month 6/5: number analyzed (Participants) | 412 | 217
  Month 6/5 | 0.8 (139.88) | 5.7 (105.08)
  Month 12/11: number analyzed (Participants) | 397 | 204
  Month 12/11 | -0.6 (123.52) | -1.2 (105.26)

22. Secondary Outcome: Change From Baseline in Renal Biomarker: Urine Retinol Binding Protein/Creatinine (Milligram Per Mole (mg/Mol))
Description: Serum samples were collected to evaluate renal specific biomarkers: urine retinol binding protein/creatinine. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: milligram per mole (mg/mol)
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 216 | 107
milligram per mole (mg/mol)
  Baseline (Day 1) | 8.6 (6.32) | 8.0 (5.75)
  Month 6/5: number analyzed (Participants) | 68 | 40
  Month 6/5 | 0.8 (6.00) | -0.8 (7.23)
  Month 12/11: number analyzed (Participants) | 91 | 50
  Month 12/11 | -0.5 (6.41) | 0.0 (4.15)

23. Secondary Outcome: Change From Baseline in Renal Biomarker: Urine Beta-2 Microglobulin/ Creatinine (Grams Per Mole (g/Mol))
Description: Serum samples were collected to evaluate renal specific biomarkers: urine beta-2 microglobulin/ creatinine. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: grams per mole (g/mol)
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 182 | 88
grams per mole (g/mol)
  Baseline (Day 1) | 0.0 (0.03) | 0.0 (0.04)
  Month 6/5: number analyzed (Participants) | 94 | 44
  Month 6/5 | 0.0 (0.03) | 0.0 (0.19)
  Month 12/11: number analyzed (Participants) | 79 | 45
  Month 12/11 | 0.0 (0.02) | 0.0 (0.04)

24. Secondary Outcome: Change From Baseline in Percentage of Participants With Metabolic Syndrome at Month 12/11
Description: Metabolic syndrome defined as cluster of conditions that occurred together increasing one's risk of heart disease, stroke and type 2 diabetes mellitus (DM). These conditions included increased blood pressure (BP), elevated blood glucose levels, excess body fat around the waist and abnormal fasting cholesterol and triglyceride (TG) levels. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. For the Q2M arm, data from the Q2M OLI participants at Month 12 visit and Q2M D2I participants at Month 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 12 visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and at Month 12/11
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 454 | 227
Percentage of participants
  Yes (Baseline) to Yes (Month 12/11) | 9 | 9
  Yes (Baseline) to No (Month 12/11) | 5 | 7
  Yes (Baseline) to Missing (Month 12/11) | 2 | 1
  No (Baseline) to Yes (Month 12/11) | 6 | 8
  No (Baseline) to No (Month 12/11) | 69 | 70
  No (Baseline) to Missing ((Month 12/11)) | 8 | 6

25. Secondary Outcome: Change From Baseline in Percentage of Participants With Metabolic Syndrome at Month 6/5
Description: Metabolic syndrome defined as cluster of conditions that occurred together increasing one's risk of heart disease, stroke and type 2 diabetes mellitus (DM). These conditions included increased blood pressure (BP), elevated blood glucose levels, excess body fat around the waist and abnormal fasting cholesterol and triglyceride (TG) levels. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. For the Q2M arm, data from the Q2M OLI participants at Month 6 visit and Q2M D2I participants at Month 5 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit.
Time Frame: Baseline (Day 1) and at month 6/5
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 454 | 227
Percentage of participants
  Yes (Baseline) to Yes (Month 6/5) | 9 | 11
  Yes (Baseline) to No (Month 6/5) | 7 | 6
  Yes (Baseline) to Missing (Month 6/5) | 1 | 0
  No (Baseline) to Yes (Month 6/5) | 5 | 10
  No (Baseline) to No (Month 6/5) | 74 | 71
  No (Baseline) to Missing (Month 6/5) | 5 | 2

26. Secondary Outcome: Change From Baseline in Homeostasis Model of Assessment-insulin Resistance (HOMA-IR)
Description: The homeostatic model assessment (HOMA) is a method used to quantify insulin resistance. HOMA-IR is calculated as fasting insulin microunits per liter (microU/L) multiplied by fasting glucose (nmol/L) divided by 22.5. Higher HOMA-IR values indicate increased insulin resistance; values <2 is generally regarded as normal. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 409 | 210
HOMA-IR score
  Baseline (Day 1) | 2.8 (4.05) | 3.1 (5.06)
  Month 6/5: number analyzed (Participants) | 348 | 191
  Month 6/5 | 0.3 (4.11) | -0.1 (5.09)
  Month 12/11: number analyzed (Participants) | 346 | 177
  Month 12/11 | 0.2 (3.99) | -0.4 (3.76)

27. Secondary Outcome: Percentage of Participants With Treatment Preference as Assessed Using Preference Questionnaire at Month 12/11 - Q2M
Description: Participants who had switched from the daily oral BIK regimen to CAB + RPV, were assessed as per the preference questionnaire every two months. There were 3 preference questions included to assess the preferred treatment 1) Long-acting injectable HIV medication, 2) Daily oral HIV medication, 3) No Preference. This endpoint was only planned to be analyzed for Q2M arm only. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit. Data represented included maintenance withdrawal or Month 12/11.
Time Frame: Up to month 12/11
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Oral lead-in Phase (OLI) | Direct to Injections (D2I)
Number analyzed (Participants) | 163 | 262
Percentage of participants
  Long-acting injectable HIV medication | 87 | 92
  Daily oral HIV medication | 7 | 4
  No Preference | 6 | 5

28. Secondary Outcome: Change From Baseline in Total Treatment Satisfaction Score Using HIV Treatment Satisfaction Status Questionnaire (HIVTSQs)
Description: The HIVTSQs total treatment satisfaction score comprised of 11 items based on HIVTSQ questionnaire each graded on a scale of 0 (very dissatisfied) to 6 (very satisfied) which were summed to produce a total score range of 0-66. Higher scores represent greater treatment satisfaction. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 446 | 222
Scores on scale
  Baseline (Day 1) | 57.88 (7.906) | 58.38 (8.229)
  Month 6/5: number analyzed (Participants) | 436 | 220
  Month 6/5 | 3.99 (9.670) | -0.66 (7.417)
  Month 12/11: number analyzed (Participants) | 410 | 213
  Month 12/11 | 4.21 (9.273) | -1.93 (8.045)

29. Secondary Outcome: Change From Baseline in Individual Item Scores Using HIVTSQs
Description: The individual item scores on HIVTSQs scale were rated on a scale of 6 (very satisfied, convenient, flexible, etc.) to -6 (very dissatisfied, inconvenient, inflexible, etc.). Higher scores represent greater satisfaction with each aspect of treatment. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline is defined as post-dose visit value minus baseline value. For the Q2M arm, data from the Q2M OLI participants at Month 6 and 12 visit and Q2M D2I participants at Month 5 and 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 6 and 12 visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: Baseline (Day 1) and up to Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 446 | 222
Scores on scale
  (Item 1=Satisfaction with current treatment), Baseline (Day 1) | 5.5 (0.86) | 5.6 (0.75)
  (Item 1=Satisfaction with current treatment), Month 6/5: number analyzed (Participants) | 436 | 220
  (Item 1=Satisfaction with current treatment), Month 6/5 | 0.1 (1.10) | -0.2 (0.91)
  (Item 1=Satisfaction with current treatment), Month 12/11: number analyzed (Participants) | 410 | 213
  (Item 1=Satisfaction with current treatment), Month 12/11 | 0.2 (1.07) | -0.3 (1.00)
  (Item 2=Controlled HIV), Baseline (Day 1) | 5.8 (0.54) | 5.8 (0.45)
  (Item 2=Controlled HIV), Month 6/5: number analyzed (Participants) | 436 | 220
  (Item 2=Controlled HIV), Month 6/5 | 0.0 (0.80) | -0.1 (0.55)
  (Item 2=Controlled HIV), Month 12/11: number analyzed (Participants) | 410 | 213
  (Item 2=Controlled HIV), Month 12/11 | 0.0 (0.70) | -0.1 (0.69)
  (Item 3=Satisfaction with side effects of present treatment), Baseline (Day 1) | 5.5 (0.91) | 5.5 (1.02)
  (Item 3=Satisfaction with side effects of present treatment), Month 6/5: number analyzed (Participants) | 436 | 220
  (Item 3=Satisfaction with side effects of present treatment), Month 6/5 | -0.3 (1.42) | 0.0 (1.21)
  (Item 3=Satisfaction with side effects of present treatment), Month 12/11: number analyzed (Participants) | 410 | 213
  (Item 3=Satisfaction with side effects of present treatment), Month 12/11 | -0.1 (1.38) | 0.0 (1.16)
  (Item 4=Satisfaction with current treatment demands), Baseline (Day 1) | 5.2 (1.16) | 5.2 (1.21)
  (Item 4=Satisfaction with current treatment demands), Month 6/5: number analyzed (Participants) | 435 | 220
  (Item 4=Satisfaction with current treatment demands), Month 6/5 | 0.4 (1.32) | -0.1 (1.28)
  (Item 4=Satisfaction with current treatment demands), Month 12/11: number analyzed (Participants) | 410 | 213
  (Item 4=Satisfaction with current treatment demands), Month 12/11 | 0.3 (1.33) | -0.2 (1.35)
  (Item 5=Treatment convenience), Baseline (Day 1) | 5.0 (1.24) | 5.2 (1.16)
  (Item 5=Treatment convenience), Month 6/5: number analyzed (Participants) | 436 | 220
  (Item 5=Treatment convenience), Month 6/5 | 0.6 (1.42) | -0.1 (1.30)
  (Item 5=Treatment convenience), Month 12/11: number analyzed (Participants) | 410 | 213
  (Item 5=Treatment convenience), Month 12/11 | 0.7 (1.43) | -0.2 (1.33)
  (Item 6=Treatment flexibility), Baseline (Day 1) | 4.7 (1.70) | 4.9 (1.55)
  (Item 6=Treatment flexibility), Month 6/5: number analyzed (Participants) | 436 | 220
  (Item 6=Treatment flexibility), Month 6/5 | 0.9 (1.77) | 0.0 (1.58)
  (Item 6=Treatment flexibility), Month 12/11: number analyzed (Participants) | 410 | 213
  (Item 6=Treatment flexibility), Month 12/11 | 0.9 (1.74) | -0.1 (1.58)
  (Item 7=Satisfaction with understanding of HIV), Baseline (Day 1) | 5.5 (0.80) | 5.5 (0.92)
  (Item 7=Satisfaction with understanding of HIV), Month 6/5: number analyzed (Participants) | 436 | 220
  (Item 7=Satisfaction with understanding of HIV), Month 6/5 | 0.2 (0.81) | 0.1 (0.75)
  (Item 7=Satisfaction with understanding of HIV), Month 12/11: number analyzed (Participants) | 410 | 213
  (Item 7=Satisfaction with understanding of HIV), Month 12/11 | 0.1 (0.86) | 0.1 (0.78)
  (Item 8=Treatment fitting in with lifestyle), Baseline (Day 1): number analyzed (Participants) | 445 | 221
  (Item 8=Treatment fitting in with lifestyle), Baseline (Day 1) | 5.0 (1.20) | 5.1 (1.11)
  (Item 8=Treatment fitting in with lifestyle), Month 6/5: number analyzed (Participants) | 434 | 218
  (Item 8=Treatment fitting in with lifestyle), Month 6/5 | 0.7 (1.36) | -0.1 (1.26)
  (Item 8=Treatment fitting in with lifestyle), Month 12/11: number analyzed (Participants) | 408 | 212
  (Item 8=Treatment fitting in with lifestyle), Month 12/11 | 0.7 (1.31) | -0.2 (1.38)
  (Item 9=Recommendation of current treatment for HIV), Baseline (Day 1): number analyzed (Participants) | 444 | 221
  (Item 9=Recommendation of current treatment for HIV), Baseline (Day 1) | 5.5 (0.86) | 5.5 (1.02)
  (Item 9=Recommendation of current treatment for HIV), Month 6/5: number analyzed (Participants) | 433 | 218
  (Item 9=Recommendation of current treatment for HIV), Month 6/5 | 0.2 (1.10) | 0.0 (1.09)
  (Item 9=Recommendation of current treatment for HIV), Month 12/11: number analyzed (Participants) | 408 | 212
  (Item 9=Recommendation of current treatment for HIV), Month 12/11 | 0.2 (1.04) | -0.1 (1.04)
  (Item 10=Satisfaction with present treatment continuation), Baseline (Day 1): number analyzed (Participants) | 445 | 221
  (Item 10=Satisfaction with present treatment continuation), Baseline (Day 1) | 4.9 (1.23) | 4.9 (1.28)
  (Item 10=Satisfaction with present treatment continuation), Month 6/5: number analyzed (Participants) | 434 | 218
  (Item 10=Satisfaction with present treatment continuation), Month 6/5 | 0.8 (1.54) | 0.0 (1.38)
  (Item 10=Satisfaction with present treatment continuation), Month 12/11: number analyzed (Participants) | 409 | 212
  (Item 10=Satisfaction with present treatment continuation), Month 12/11 | 0.9 (1.49) | -0.2 (1.45)
  (Item 11=Ease or difficulty with current treatment), Baseline (Day 1): number analyzed (Participants) | 445 | 221
  (Item 11=Ease or difficulty with current treatment), Baseline (Day 1) | 5.2 (1.10) | 5.3 (1.06)
  (Item 11=Ease or difficulty with current treatment), Month 6/5: number analyzed (Participants) | 434 | 218
  (Item 11=Ease or difficulty with current treatment), Month 6/5 | 0.5 (1.34) | -0.2 (1.20)
  (Item 11=Ease or difficulty with current treatment), Month 12/11: number analyzed (Participants) | 409 | 212
  (Item 11=Ease or difficulty with current treatment), Month 12/11 | 0.5 (1.34) | -0.3 (1.13)
  (Item 12=Satisfaction with amount of discomfort/pain with current treatment), Baseline (Day 1): number analyzed (Participants) | 445 | 221
  (Item 12=Satisfaction with amount of discomfort/pain with current treatment), Baseline (Day 1) | 5.5 (1.02) | 5.6 (0.94)
  (Item 12=Satisfaction with amount of discomfort/pain with current treatment), Month 6/5: number analyzed (Participants) | 434 | 218
  (Item 12=Satisfaction with amount of discomfort/pain with current treatment), Month 6/5 | -0.6 (1.64) | -0.1 (0.93)
  (Item 12=Satisfaction with amount of discomfort/pain with current treatment), Month 12/11: number analyzed (Participants) | 409 | 212
  (Item 12=Satisfaction with amount of discomfort/pain with current treatment), Month 12/11 | -0.5 (1.54) | -0.2 (1.09)

30. Secondary Outcome: HIV Treatment Satisfaction Change Questionnaire (HIVTSQc) Total Score at Month 12/11
Description: HIV treatment satisfaction change questionnaire (HIVTSQc) total Score is computed with items 1-11 which were summed to produce a total score range of -33 to 33. Higher score indicated greater improvement in the satisfaction with the treatment and lower score indicated greater deterioration in treatment satisfaction. A score of 0 represents no change. For the Q2M arm, data from the Q2M OLI participants at Month 12 visit and Q2M D2I participants at Month 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 12 visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: At Month 12/11
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 426 | 214
Scores on scale | 26.97 (10.135) | 16.89 (14.299)

31. Secondary Outcome: Individual Item Scores of HIVTSQc at Month 12/11
Description: Individual item scores were rated on a scale of +3 (much more satisfied', 'much more convenient', 'much more flexible') to -3 (much less satisfied', 'much less convenient', 'much less flexible'). Higher score indicates greater improvement, and lower score indicates greater deterioration in satisfaction with each aspect of treatment. A score of 0 represents no change. For the Q2M arm, data from the Q2M OLI participants at Month 12 visit and Q2M D2I participants at Month 11 visit were combined as the study objective was to demonstrate the non-inferior antiviral activity of (Q2M) (OLI+ D2I combined) compared to BIK. For BIK arm, data was collected at month 12 visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: At Month 12/11
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Q2M (OLI + D2I) | Biktarvy (BIK)
Number analyzed (Participants) | 427 | 214
Scores on scale
  Item 1=Satisfaction with current treatment | 2.56 (1.043) | 1.60 (1.417)
  Item 2=Controlled HIV: number analyzed (Participants) | 425 | 214
  Item 2=Controlled HIV | 2.47 (1.086) | 1.88 (1.375)
  Item 3=Satisfaction with side effects of present treatment: number analyzed (Participants) | 426 | 214
  Item 3=Satisfaction with side effects of present treatment | 2.10 (1.388) | 1.63 (1.463)
  Item 4=Satisfaction with current treatment demands: number analyzed (Participants) | 426 | 214
  Item 4=Satisfaction with current treatment demands | 2.41 (1.109) | 1.42 (1.560)
  Item 5=Treatment convenience: number analyzed (Participants) | 426 | 214
  Item 5=Treatment convenience | 2.50 (1.070) | 1.38 (1.520)
  Item 6=Treatment flexibility: number analyzed (Participants) | 426 | 214
  Item 6=Treatment flexibility | 2.41 (1.138) | 1.24 (1.591)
  Item 7=Satisfaction with understanding of HIV: number analyzed (Participants) | 425 | 214
  Item 7=Satisfaction with understanding of HIV | 2.35 (1.065) | 1.94 (1.297)
  Item 8=Treatment fitting in with lifestyle: number analyzed (Participants) | 425 | 214
  Item 8=Treatment fitting in with lifestyle | 2.56 (0.994) | 1.43 (1.489)
  Item 9=Recommendation of current treatment for HIV: number analyzed (Participants) | 425 | 214
  Item 9=Recommendation of current treatment for HIV | 2.61 (1.065) | 1.73 (1.467)
  Item 10=Satisfaction with present treatment continuation: number analyzed (Participants) | 424 | 214
  Item 10=Satisfaction with present treatment continuation | 2.58 (1.093) | 1.22 (1.602)
  Item 11=Ease or difficulty with current treatment: number analyzed (Participants) | 425 | 214
  Item 11=Ease or difficulty with current treatment | 2.46 (1.107) | 1.43 (1.542)
  Item 12=Satisfaction with amount of discomfort/pain with current treatment: number analyzed (Participants) | 425 | 214
  Item 12=Satisfaction with amount of discomfort/pain with current treatment | 1.85 (1.530) | 1.64 (1.465)

32. Secondary Outcome: Change From Month 2/1 in Dimension Scores Using Perception of Injection (PIN) Questionnaire - Q2M
Description: The PIN questionnaire was used to explore the dimension scores based on 4 dimensions including acceptance of injection site reactions (ISRs), Bother from ISRs, Leg movement and Sleep categories. Domain scores were calculated as a mean of all items with the domain. The PIN response options range from 1 (totally acceptable) to 5 (not at all acceptable). This endpoint was only planned to be analyzed for Q2M arm. Month 2/1 refers to the Month 2 (OLI and BIK) visit/Month 1 (DTI) visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: From Month 2/1 up to Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Oral lead-in Phase (OLI) | Direct to Injections (D2I)
Number analyzed (Participants) | 163 | 271
Scores on scale
  Bother of ISRs, Month 2/1 | 1.58 (0.568) | 1.60 (0.583)
  Bother of ISRs, Month 6/5: number analyzed (Participants) | 160 | 263
  Bother of ISRs, Month 6/5 | 0.01 (0.528) | -0.03 (0.590)
  Bother of ISRs, Month 12/11: number analyzed (Participants) | 152 | 255
  Bother of ISRs, Month 12/11 | 0.08 (0.594) | -0.04 (0.583)
  Leg Movement, Month 2/1: number analyzed (Participants) | 163 | 270
  Leg Movement, Month 2/1 | 1.93 (1.013) | 1.83 (0.913)
  Leg Movement, Month 6/5: number analyzed (Participants) | 160 | 262
  Leg Movement, Month 6/5 | -0.14 (0.779) | -0.22 (0.868)
  Leg Movement, Month 12/11: number analyzed (Participants) | 152 | 254
  Leg Movement, Month 12/11 | -0.18 (0.859) | -0.24 (0.817)
  Sleep, Month 2/1: number analyzed (Participants) | 163 | 270
  Sleep, Month 2/1 | 1.83 (0.936) | 1.87 (0.965)
  Sleep, Month 6/5: number analyzed (Participants) | 160 | 262
  Sleep, Month 6/5 | -0.01 (0.915) | -0.16 (0.869)
  Sleep, Month 12/11: number analyzed (Participants) | 152 | 254
  Sleep, Month 12/11 | -0.07 (0.948) | -0.17 (0.870)
  Acceptance, Month 2/1 | 2.02 (1.017) | 2.05 (0.949)
  Acceptance, Month 6/5: number analyzed (Participants) | 160 | 263
  Acceptance, Month 6/5 | -0.14 (0.906) | -0.13 (0.879)
  Acceptance, Month 12/11: number analyzed (Participants) | 152 | 255
  Acceptance, Month 12/11 | -0.20 (0.873) | -0.26 (0.856)

33. Secondary Outcome: Change From Month 2/1 in Individual Item Scores Using PIN Questionnaire- Q2M
Description: The PIN questionnaire was used to explore the individual item scores based on anxiety before, pain, satisfaction, anxiety after and willingness categories. The items in the scale are rated on a 5-point scale and questions are phrased in such a way as to ensure that 1 is very dissatisfied and 5 was very satisfied. This endpoint was only planned to be analyzed for Q2M arm. Month 2/1 refers to the Month 2 (OLI and BIK) visit/Month 1 (DTI) visit. Month 6/5 refers to the Month 6 (OLI and BIK) visit/Month 5 (DTI) visit. Month 12/11 refers to the Month 12 (OLI and BIK) visit/Month 11 (DTI) visit.
Time Frame: From Month 2/1 up to Month 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Oral lead-in Phase (OLI) | Direct to Injections (D2I)
Number analyzed (Participants) | 163 | 271
Scores on scale
  Anxiety Before, Month 2/1 | 1.9 (1.02) | 1.9 (1.02)
  Anxiety Before, Month 6/5: number analyzed (Participants) | 160 | 263
  Anxiety Before, Month 6/5 | -0.14 (1.021) | -0.22 (1.000)
  Anxiety Before, Month 12/11: number analyzed (Participants) | 152 | 255
  Anxiety Before, Month 12/11 | -0.28 (0.973) | -0.22 (0.914)
  Pain, Month 2/1 | 1.8 (0.88) | 2.0 (0.93)
  Pain, Month 6/5: number analyzed (Participants) | 160 | 263
  Pain, Month 6/5 | 0.09 (0.907) | -0.03 (0.935)
  Pain, Month 12/11: number analyzed (Participants) | 152 | 255
  Pain, Month 12/11 | 0.13 (0.995) | 0.02 (0.943)
  Satisfaction, Month 2/1 | 1.7 (0.90) | 1.6 (0.81)
  Satisfaction, Month 6/5: number analyzed (Participants) | 160 | 263
  Satisfaction, Month 6/5 | -0.06 (0.837) | 0.00 (0.867)
  Satisfaction, Month 12/11: number analyzed (Participants) | 152 | 255
  Satisfaction, Month 12/11 | -0.12 (0.861) | -0.11 (0.830)
  Anxiety After, Month 2/1 | 1.8 (1.12) | 1.7 (0.96)
  Anxiety After, Month 6/5: number analyzed (Participants) | 160 | 263
  Anxiety After, Month 6/5 | -0.14 (0.994) | -0.04 (0.916)
  Anxiety After, Month 12/11: number analyzed (Participants) | 152 | 255
  Anxiety After, Month 12/11 | -0.24 (0.947) | -0.16 (0.850)
  Willingness, Month 2/1: number analyzed (Participants) | 162 | 271
  Willingness, Month 2/1 | 1.4 (0.76) | 1.4 (0.78)
  Willingness, Month 6/5: number analyzed (Participants) | 157 | 263
  Willingness, Month 6/5 | 0.01 (0.716) | -0.08 (0.794)
  Willingness, Month 12/11: number analyzed (Participants) | 151 | 254
  Willingness, Month 12/11 | -0.01 (0.744) | -0.10 (0.742)

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to end of Extension Phase (approximately Month 27).
Description: AEs are reported based on Safety set population, which included all randomized participants who received at least one dose of study drug, based on the study phase they were included in. The Safety set included all participants irrespective of eligibility criteria violation and GCP non-compliance, since they received at least a study intervention dose.
Arm/Group | Oral lead-in Phase (OLI) | Direct to Injections (D2I) | Biktarvy (BIK) | Switch Q2M Group
All-Cause Mortality (participants affected / at risk) | 0/175 | 0/279 | 1/227 | 1/145
Serious Adverse Events (participants affected / at risk) | 11/175 | 10/279 | 15/227 | 5/145
Other Adverse Events (participants affected / at risk) | 156/175 | 257/279 | 77/227 | 76/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral lead-in Phase (OLI) (N=175) | Direct to Injections (D2I) (N=279) | Biktarvy (BIK) (N=227) | Switch Q2M Group (N=145)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex meningoencephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorectal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral lead-in Phase (OLI) (N=175) | Direct to Injections (D2I) (N=279) | Biktarvy (BIK) (N=227) | Switch Q2M Group (N=145)
Injection site pain (General disorders) | 106 (106) | 182 (182) | 1 (2) | 55 (55)
Injection site nodule (General disorders) | 17 (17) | 26 (26) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 15 (15) | 27 (27) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 10 (10) | 26 (26) | 8 (8) | 0 (0)
Injection site discomfort (General disorders) | 17 (17) | 26 (26) | 0 (0) | 0 (0)
Fatigue (General disorders) | 17 (17) | 14 (14) | 6 (7) | 0 (0)
Injection site induration (General disorders) | 20 (20) | 17 (17) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 34 (34) | 50 (50) | 38 (38) | 21 (21)
Nasopharyngitis (Infections and infestations) | 8 (8) | 25 (25) | 10 (13) | 0 (0)
Syphilis (Infections and infestations) | 8 (8) | 23 (23) | 9 (10) | 0 (0)
Headache (Nervous system disorders) | 17 (17) | 35 (35) | 12 (12) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 21 (21) | 9 (9) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 17 (17) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 16 (16) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT04542070/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT04542070/SAP_001.pdf